CLINICAL TRIAL: NCT01545999
Title: Paired Associative Stimulation in the Dorsolateral Prefrontal Cortex in Patients With Schizophrenia: a Combined Transcranial Magnetic Stimulation and Electroencephalography Study Across the Life Span
Brief Title: Paired Associative Stimulation in the Dorsolateral Prefrontal Cortex in Patients With Schizophrenia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Tarek Rajji, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #165/2009-04
Record Dates: First submitted 2012-01-17; First posted 2012-03-07 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia
Keywords: Transcranial Magnetic Stimulation (TMS); Dorsolateral Prefrontal Cortex (DLPFC); Schizophrenia; Working Memory; Paired Associative Stimulation (PAS); Electroencephalography (EEG); Cognition
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PAS 25 (Active Comparator): In humans, paired associative stimulation (PAS-25) is a transcranial magnetic stimulation (TMS) protocol that has been shown to result in LTP-like plasticity (PAS-LTP) in the motor cortex (M1). PAS-LTP has been shown to be dependent on the NMDAR and to correlate significantly with performance on a motor learning task.
  Interventions: Other: Brain Stimulation via Transcranial Magnetic Stimulation
- PAS 100 (Sham Comparator): To control for non-specific effects of PAS protocol, the investigators will use a modified PAS protocol (PAS-100) that does not result in any neurophysiologic effects. Patients with schizophrenia and healthy controls will be assessed first with the N-back task and then randomized
  Interventions: Other: Brain Stimulation via Transcranial Magnetic Stimulation

INTERVENTIONS:
Other: Brain Stimulation via Transcranial Magnetic Stimulation — PAS-25 will consist of 180 PNS delivered to right median nerve, each paired with a single TMS pulse delivered over left DLPFC with an interstimulus interval of 25 ms. This ISI was designed to generate approximately synchronous arrival of both inputs in M1 and was reported to markedly enhance TMS-induced MEP following PAS-25.
  Patients with schizophrenia will be asked to continue with a 2-week course (5 days/week) of daily PAS-25 or PAS-100 to assess potential of a repetitive course of PAS-25 on enhancing working memory in patients with Schizophrenia. One and seven days after the 2-week course PAS-25 or PAS-100, patients with schizophrenia will be assessed with the N-back task.

SUMMARY:
The purpose of this study is to

1. assess the effect of PAS in schizophrenia in the dorsolateral prefrontal cortex (DLPFC)
2. assess the effect of PAS induced long-term potentiation (LTP) on the performance of patients with schizophrenia on a cognitive task related to DLFPC.

DETAILED DESCRIPTION:
Neuroplasticity refers to changes in the strength of communication between different neurons. Long-term potentiation (LTP) is one form of neuroplasticity and refers to the strengthening of such communication. LTP is believed to be a cellular substrate of learning and memory. Paired associative stimulation (PAS) is a transcranial magnetic stimulation (TMS) paradigm that is believed to induce LTP in human subjects. However, its effects have been shown to be minimal in patients with schizophrenia suggesting impaired LTP in schizophrenia. The lack of PAS effect in schizophrenia has been observed in the motor cortex (M1). Thus, the investigators propose to assess the effect of PAS in schizophrenia in the dorsolateral prefrontal cortex (DLPFC), an area of the brain that is especially relevant to learning and memory, and to the pathology in schizophrenia. The investigators also propose to assess the effect of PAS induced LTP on the performance of patients with schizophrenia on a cognitive task that is related to DLFPC.

Hypothesis 1: Patients with schizophrenia will have reduced PAS-LTP in DLPFC in comparison with healthy controls.

Hypothesis 2a: PAS-LTP in patients with schizophrenia and healthy controls randomized to PAS-25 and PAS-100 will correlate with performance on the N-back task at baseline (pre-PAS).

Hypothesis 2b: Healthy controls randomized to PAS-25 will perform better after one session of PAS-25 on the 1- and 7-day N-back task compared to healthy controls randomized to PAS-100.

Hypothesis 2c: Among healthy controls randomized to PAS-25, the magnitude of improvement on the 1- and 7-day N-back task (compared to pre-PAS) that is in excess of the magnitude of improvement on the 1- and 7-day N-back task among subjects randomized to PAS-100 will correlate with the degree of PAS-LTP.

Hypothesis 3a: Patients with schizophrenia who are randomized to receive a 2-week course of PAS-25 will have improved PAS-LTP in DLPFC compared to patients with schizophrenia randomized to 2-week course of PAS-100.

Hypothesis 3b: Patients with schizophrenia who are randomized to receive a 2-week course of PAS-25 will have improved performance on the N-back working memory task compared to patients with schizophrenia randomized to 2-week PAS-100 at 1- and 7-day post-PAS course N-back.

Hypothesis 3c: Patients with schizophrenia who are randomized to receive a 2-week course of PAS-25 will have increased DLPFC cortical thickness compared to patients with schizophrenia randomized to 2-week PAS-100.

Hypothesis 4: Among patients with schizophrenia and healthy controls, PAS-LTP will decrease with age, and the decrease will be more pronounced in healthy controls than in patients.

ELIGIBILITY:
Inclusion Criteria for patients:

* Age 18 or above
* All races and ethnicities.
* Females and males.
* Meet DSM-IV TR criteria for a current diagnosis of schizophrenia or schizoaffective disorder.
* Clinically stable as operationalized by (1) either having not been hospitalized within 3 months or having been hospitalized for 3 months or more prior to assessment, and (2) having had no change in antipsychotic medication dosage within the 4 weeks prior to assessment.
* Willingness and ability to speak English
* Willingness to provide informed consent
* Corrected visual ability that enables reading of newspaper headlines and corrected hearing capacity that is adequate to respond to a raised conversational voice.

Exclusion Criteria for patients:

* Meets criteria for a cognitive disorder secondary to a neurological or other medical disorder affecting the central nervous system (for example, multiple sclerosis, history of traumatic brain injury, stroke, untreated hypothyroidism).
* Mini Mental Status Examination score of 17 and less because a subject with a very low MMSE score is unlikely to be able to compete the NP battery.
* Diagnosis of bipolar disorder or current major depressive episode.
* Meets diagnostic criteria for current alcohol or other drug dependence within 6 months of testing
* Electroconvulsive Therapy (ECT) within 6 months of testing.
* Left handedness.
* Incompetency to consent

Inclusion Criteria for controls:

* Age 18 or above
* Willingness and ability to speak English
* Willingness to provide informed consent
* Corrected visual ability that enables reading of newspaper headlines and corrected hearing capacity that is adequate to respond to a raised conversational voice.

Exclusion Criteria for controls:

* DSM IV TR psychiatric diagnosis except for simple phobias or an adjustment disorder.
* Other neurological disorder affecting central nervous system.
* Psychotropic medication except for sedative /hypnotics at a stable dose for at least 4 weeks.
* Family history of a primary psychotic disorder in a first-degree relative.
* Left handedness.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2012-03; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in working memory | 1 day and 7 days post N-back task
  The N-Back is a working memory task where the subject is presented with a sequence of stimuli (letters). The task consists of indicating when the current stimulus matches the one from n steps earlier in the sequence. The load factor n can be adjusted to make the task more or less difficult. Subjects are required to complete the 0, 1, 2 and 3 back at baseline, 1 day post PAS delivery and 7 days post PAS.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek K Rajji, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching — http://www.camh.net/research